CLINICAL TRIAL: NCT04908800
Title: A First-in-Human, Phase I, Double-blind, Placebo-controlled, Single and Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of KRP-A218 in Healthy Subjects, Including Food-Effect and Drug-drug Interaction With Itraconazole
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of KRP-A218 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: KRPA218-T101
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Results first posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2023-03

CONDITIONS: Healthy
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A single ascending dose (SAD) and Part B multiple ascending dose (MAD): KRP-A218 (Experimental): Administration Route: Oral
  Interventions: Drug: KRP-A218
- Part A (SAD) and Part B (MAD): Placebo (Placebo Comparator): Administration Route: Oral
  Interventions: Drug: Placebo
- Part C drug-drug interaction (DDI): KRP-A218 and itraconazole (Experimental): Administration Route: Oral
  Interventions: Drug: KRP-A218; Drug: itraconazole

INTERVENTIONS:
Drug: KRP-A218 — KRP-A218 tablet
  Arms: Part A single ascending dose (SAD) and Part B multiple ascending dose (MAD): KRP-A218; Part C drug-drug interaction (DDI): KRP-A218 and itraconazole
Drug: Placebo — Placebo tablet
  Arms: Part A (SAD) and Part B (MAD): Placebo
Drug: itraconazole — 10 mg/mL oral solution
  Other Names: Sporanox
  Arms: Part C drug-drug interaction (DDI): KRP-A218 and itraconazole

SUMMARY:
This first-in-human study has three parts. In Parts A and B, the safety, tolerability, and pharmacokinetics (PK) will be evaluated following administration of single and multiple doses of KRP-A218, including food-effect. In Part C, the drug-drug interaction (DDI) with itraconazole will be evaluated.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female adults, between 20 and 55 years of age, inclusive.
* Body weight ≥50 kg, with body mass index (BMI) between 18.0 and 30.0 kg/m^2, inclusive.
* In good health, at Screening or Day -1 as assessed by the Investigator.
* Females will not be pregnant or lactating, and females of childbearing potential will agree to use contraception and to not donate eggs (ova, oocytes). Males will agree to use contraception and to not donate sperm.
* Able to comprehend and willing to sign an informed consent form (ICF) and to abide by the study restrictions.

Key Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, haematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing.
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing.
* Use or intend to use any prescription medications/products within 14 days or 5 half-lives (whichever is longer) prior to dosing, unless deemed acceptable by the Investigator.
* Use or intend to use slow release medications/products considered to still be active within 14 days prior to dosing, unless deemed acceptable by the Investigator.
* Use or intend to use any nonprescription medications/products including vitamins, minerals, and phytotherapeutic/herbal/plant derived preparations within 7 days prior to dosing, unless deemed acceptable by the Investigator.
* Use of tobacco or nicotine-containing products within 3 months prior to Day -1, or positive cotinine test at screening or Day -1.
* Ingestion of poppy seed-, Seville orange-, or grapefruit-containing foods or beverages within 7 days prior to Day -1.
* Consumption of caffeine- or xanthine-containing foods and beverages within 36 hours prior to Day -1.
* Participation in strenuous exercised within 7 days prior to Day -1.
* Receipt of blood products within 2 months prior to Day -1.
* Donation of blood from 3 months prior to screening, plasma from 2 weeks prior to screening, or platelets from 6 weeks prior to screening.
* Poor peripheral venous access.
* Have previously completed or withdrawn from this study or have previously received the investigational medicinal product (IMP).
* Subject is, in the opinion of the Investigator, unlikely to comply with the protocol or unsuitable to participate in this study for any reason.

Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoji Mimaki, Study Chair — Kyorin Pharmaceutical Co.,Ltd
Locations (1):
- Labcorp Clinical Research, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A: Placebo: Single ascending dose study.
  Participants received a single order dose of placebo with approximately 240 mL of room temperature water after an overnight fast of at least 10 hours.
  For those randomized to the Fasted/Fed group, on Day 1, Treatment Period 2, male participants also received a single order dose of placebo 30 minutes after starting a high-fat breakfast.
- Part A: 1 mg KRP-A218 (Fasted Male): Single ascending dose study.
  Participants received a single order dose of 1 mg KRP-A218 with approximately 240 mL of room temperature water after an overnight fast of at least 10 hours.
- Part A: 3 mg KRP-A218 (Fasted/Fed Male): Single ascending dose study.
  On Day 1, Treatment Period 1, male participants received a single order dose of 3 mg KRP-A218 after an overnight fast of at least 10 hours.
  On Day 1, Treatment Period 2, male participants received a single order dose of 3 mg KRP-A218 30 minutes after starting a high-fat breakfast.
- Part A: 3 mg KRP-A218 (Fasted Female): Single ascending dose study.
  Female participants received a single order dose of 3 mg KRP-A218 with approximately 240 mL of room temperature water after an overnight fast of at least 10 hours.
- Part A: 6 mg KRP-A218 (Fasted Male): Single ascending dose study.
  Male participants received a single order dose of 6 mg KRP-A218 with approximately 240 mL of room temperature water after an overnight fast of at least 10 hours.
- Part A: 12 mg KRP-A218 (Fasted Male): Single ascending dose study.
  Male participants received a single order dose of 12 mg KRP-A218 with approximately 240 mL of room temperature water after an overnight fast of at least 10 hours.
- Part A: 21 mg KRP-A218 (Fasted Male): Single ascending dose study.
  Male participants received a single order dose of 21 mg KRP-A218 with approximately 240 mL of room temperature water after an overnight fast of at least 10 hours.
- Part B: Placebo: Multiple ascending dose study.
  Participants received once daily oral doses of placebo from Days 1 to 14. Each dose was administered with approximately 240 mL of room temperature water.
- Part B: 2 mg KRP-A218: Multiple ascending dose study.
  Participants received once daily oral doses of 2 mg KRP-A218 from Days 1 to 14. Each dose was administered with approximately 240 mL of room temperature water.
- Part B: 4 mg KRP-A218: Multiple ascending dose study.
  Participants received once daily oral doses of 4 mg KRP-A218 from Days 1 to 14. Each dose was administered with approximately 240 mL of room temperature water.
- Part B: 8 mg KRP-A218: Multiple ascending dose study.
  Participants received once daily oral doses of 8 mg KRP-A218 from Days 1 to 14. Each dose was administered with approximately 240 mL of room temperature water.
- Part B: 11 mg KRP-A218: Multiple ascending dose study.
  Participants received once daily oral doses of 11 mg KRP-A218 from Days 1 to 14. Each dose was administered with approximately 240 mL of room temperature water.
- Part C: Drug-drug Interaction Study: Days 1 and 11: single oral dose of 1 mg KRP-A218 (with approximately 240 mL of room temperature water), in the fasted state.
  Day 4: 2 × single oral doses of 200 mg itraconazole solution (10 mg/mL) administered with no additional water, approximately 12 hours apart, in the fasted state.
  Days 5 to 13: single oral doses of 200 mg itraconazole, solution (10 mg/mL) administered with no additional water, in the fasted state.
Period: Overall Study
Arm/Group | Part A: Placebo | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted/Fed Male) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male) | Part B: Placebo | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218 | Part C: Drug-drug Interaction Study
Started | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 8 | 12
Completed | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 7 | 8 | 12
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted/Fed Male) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male) | Part B: Placebo | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218 | Part C: Drug-drug Interaction Study | Total
Number analyzed (Participants) | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 8 | 12 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (6.43) | 27.4 (2.41) | 35.0 (12.68) | 36.3 (11.91) | 38.8 (9.39) | 31.0 (6.13) | 30.8 (4.71) | 36.5 (13.78) | 32.3 (9.77) | 38.4 (10.77) | 37.5 (9.96) | 31.9 (9.48) | 36.4 (11.01) | 34.3 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8
  Male | 10 | 5 | 6 | 0 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 8 | 12 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 8 | 8 | 8 | 8 | 8 | 12 | 99
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 8
  White | 10 | 5 | 5 | 4 | 6 | 4 | 5 | 6 | 7 | 7 | 7 | 7 | 12 | 85
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimetres] | 174.42 (9.549) | 180.80 (4.970) | 170.00 (3.347) | 165.33 (4.082) | 180.33 (7.394) | 180.33 (2.503) | 181.00 (7.239) | 174.13 (3.796) | 180.63 (5.449) | 182.13 (4.121) | 174.63 (8.634) | 175.63 (5.975) | 180.25 (7.275) | 176.96 (7.593)
Body Weight [Mean (Standard Deviation); unit: kilograms] | 74.44 (10.453) | 82.08 (12.815) | 72.50 (9.134) | 65.23 (8.138) | 85.80 (8.734) | 83.20 (7.654) | 82.37 (11.934) | 74.34 (7.558) | 82.01 (10.405) | 83.29 (8.061) | 74.75 (14.155) | 81.33 (11.106) | 79.20 (7.228) | 78.33 (10.653)
Body Mass Index [Mean (Standard Deviation); unit: kilograms/metres squared] | 24.43 (2.411) | 25.00 (2.769) | 25.12 (3.589) | 23.90 (3.239) | 26.35 (1.866) | 25.55 (1.981) | 25.03 (2.166) | 24.48 (1.855) | 25.06 (2.304) | 25.15 (2.718) | 24.36 (3.225) | 26.39 (3.321) | 24.38 (1.847) | 24.95 (2.519)

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Adverse Events
Description: A treatment-emergent adverse event (TEAE) was defined as an adverse event that started during or after the first dose, or started prior to the first dose and increased in severity after the first dose.
  Where a subject experienced multiple TEAEs with the same preferred term for the same treatment, this was counted as 1 TEAE for that treatment under the maximum severity recorded.
Time Frame: Screening to follow-up (Approximately 6 weeks)
Population: Safety population
Measure: Number; unit: participants
Groups:
- Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1); Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2): Single ascending dose study.
  On Day 1, Treatment Period 1, male participants received a single order dose of 3 mg KRP-A218 after an overnight fast of at least 10 hours.
  On Day 1, Treatment Period 2, male participants received a single order dose of 3 mg KRP-A218 30 minutes after starting a high-fat breakfast.
Arm/Group | Part A: Placebo | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 12 | 5 | 6 | 6 | 6 | 6 | 6 | 6
participants
  Overall TEAEs | 4 | 3 | 4 | 3 | 2 | 2 | 3 | 2
  Serious TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs Leading to Discontinuation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  TEAEs Leading to Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Part B: Number of Participants With Adverse Events
Description: as for outcome 1
Time Frame: Screening to follow-up (Approximately 8 weeks)
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Part B: Placebo | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
participants
  Overall TEAEs | 6 | 3 | 7 | 5 | 5
  Serious TEAEs | 0 | 0 | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0 | 1 | 0
  TEAEs leading to death | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part C: Area Under Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-infinity)
Description: The area under concentration-time curve from time 0 extrapolated to infinity (AUC0-infinity) following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Population: Pharmacokinetic Population)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone: Drug-drug Interaction Study: Single dose of 1 mg KRP-A218 on Day 1
- Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole: Drug-drug Interaction Study: Single dose of 1 mg KRP-A218 + 200 mg Itraconazole (QD) on Day 11
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
ng*h/mL | 191 (23.9) | 360 (25.0)
Statistical Analysis 1: Comparison: Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone vs Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.88, 90% CI 2-sided [1.74 to 2.04] — Data were analyzed using a mixed model which included actual treatment as fixed effect and participant as a random effect. Within-subject coefficient of variation was 10.7

4. Primary Outcome: Part C: Area Under Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast)
Description: The area under concentration-time curve from time 0 extrapolated to last quantifiable concentration following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
ng*h/mL | 182 (22.8) | 306 (23.5)
Statistical Analysis 1: Comparison: Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone vs Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.68, 90% CI 2-sided [1.57 to 1.79] — Data were analyzed using a mixed model which included actual treatment as fixed effect and participant as a random effect. Within-subject coefficient of variation was 9.01

5. Primary Outcome: Part C: Maximum Observed Concentration (Cmax)
Description: The maximum observed concentration following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
ng/mL | 10.7 (20.3) | 12.2 (20.9)
Statistical Analysis 1: Comparison: Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone vs Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.15, 90% CI 2-sided [1.09 to 1.21] — Data were analyzed using a mixed model which included actual treatment as fixed effect and participant as a random effect. Within-subject coefficient of variation was 7.18

6. Primary Outcome: Part C: Time of the Maximum Observed Concentration (Tmax)
Description: The time of the maximum observed concentration following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: hours
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
hours | 3.00 [2.00 to 4.00] | 2.00 [1.50 to 4.00]

7. Primary Outcome: Part C: Apparent Terminal Elimination Half-life (t1/2)
Description: The apparent terminal elimination half-life following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
hours | 15.9 (10.1) | 26.5 (15.5)

8. Primary Outcome: Part C: Apparent Total Clearance (CL/F)
Description: The apparent total clearance following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter Per Hour
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
Liter Per Hour | 5.24 (23.9) | 2.78 (25.0)

9. Primary Outcome: Part C: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Description: The apparent volume of distribution during the terminal phase following Oral Dose Administration of KRP-A218 Alone and in Combination with Itraconazole
Time Frame: Days 1 to 11
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12
liters | 120 (17.6) | 106 (23.8)

10. Secondary Outcome: Part A: Area Under Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-infinity)
Description: Area under concentration-time curve from time 0 extrapolated to infinity following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 210 (18.8) | 600 (43.2) | 607 (36.9) | 634 (18.0) | 1230 (28.3) | 2600 (23.9) | 3810 (17.9)
Statistical Analysis 1: Comparison: Part A: 1 mg KRP-A218 (Fasted Male) vs Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fasted Female) vs Part A: 6 mg KRP-A218 (Fasted Male) vs Part A: 12 mg KRP-A218 (Fasted Male) vs Part A: 21 mg KRP-A218 (Fasted Male); Dose Proportionality Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Slope = 0.971, 95% CI 2-sided [0.882 to 1.06] — Between-subject geometric coefficient of variation was 26.1. Data were analyzed using a power model
Statistical Analysis 2: Comparison: Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2); Food Effect Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.01, 95% CI 2-sided [0.926 to 1.11] — Geometric least squares mean was 600 (fasted) and 607 (fed). Within-subject coefficient of variation was 6.01. Data were analyzed using mixed model which included actual treatment as fixed effect and participant as a random effect
Statistical Analysis 3: Comparison: Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fasted Female); Sex Effect Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.06, 95% CI 2-sided [0.701 to 1.59] — Geometric least squares mean was 600 (fasted male) and 634 (fasted female). Between subject coefficient of variation was 32.7. Data were analyzed using an ANOVA model which included actual treatment as a factor

11. Secondary Outcome: Part A: Area Under Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast)
Description: Area under curve from time 0 to the time of the last quantifiable concentration following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng*h/mL | 198 (18.4) | 575 (40.4) | 578 (33.3) | 600 (18.4) | 1160 (28.4) | 2490 (24.0) | 3680 (17.5)
Statistical Analysis 1: Comparison: Part A: 1 mg KRP-A218 (Fasted Male) vs Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fasted Female) vs Part A: 6 mg KRP-A218 (Fasted Male) vs Part A: 12 mg KRP-A218 (Fasted Male) vs Part A: 21 mg KRP-A218 (Fasted Male); Dose Proportionality Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Slope = 0.977, 95% CI 2-sided [0.891 to 1.06] — Between-subject geometric coefficient of variation was 25.4. Data were analyzed using a power model
Statistical Analysis 2: Comparison: Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2); Food Effect Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.00, 95% CI 2-sided [0.905 to 1.12] — Geometric least squares mean was 575 (fasted) and 578 (fed). Within-subject coefficient of variation was 7.05. Data were analyzed using mixed model which included actual treatment as fixed effect and participant as a random effect
Statistical Analysis 3: Comparison: Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fasted Female); Sex Effect Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.04, 95% CI 2-sided [0.707 to 1.54] — Geometric least squares mean was 575 (fasted male) and 600 (fasted female). Between subject coefficient of variation was 31.1. Data were analyzed using an ANOVA model which included actual treatment as a factor

12. Secondary Outcome: Part A: Maximum Observed Concentration (Cmax)
Description: Maximum observed concentration following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 11.9 (30.3) | 31.6 (27.7) | 30.0 (16.6) | 38.8 (14.6) | 60.3 (26.5) | 146 (16.5) | 236 (15.9)
Statistical Analysis 1: Comparison: Part A: 1 mg KRP-A218 (Fasted Male) vs Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fasted Female) vs Part A: 6 mg KRP-A218 (Fasted Male) vs Part A: 12 mg KRP-A218 (Fasted Male) vs Part A: 21 mg KRP-A218 (Fasted Male); Dose Proportionality Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Slope = 0.989, 95% CI 2-sided [0.909 to 1.07] — Between-subject geometric coefficient of variation was 23.0. Data were analyzed using a power model
Statistical Analysis 2: Comparison: Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2); Food Effect Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 0.948, 95% CI 2-sided [0.824 to 1.09] — Geometric least squares mean was 31.6 (fasted) and 30.0 (fed). Within-subject coefficient of variation was 9.44. Data were analyzed using mixed model which included actual treatment as fixed effect and participant as a random effect
Statistical Analysis 3: Comparison: Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) vs Part A: 3 mg KRP-A218 (Fasted Female); Sex Effect Assessment; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Ratio of geometric least squares mean = 1.23, 95% CI 2-sided [0.928 to 1.62] — Geometric least squares mean was 31.6 (fasted male) and 38.8 (fasted female). Between subject coefficient of variation was 22.0. Data were analyzed using an ANOVA model which included actual treatment as a factor

13. Secondary Outcome: Part A: Time of the Maximum Observed Concentration (Tmax)
Description: Time of the maximum observed concentration following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: hours
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
hours | 3.00 [2.00 to 4.00] | 4.00 [2.02 to 4.00] | 3.50 [1.50 to 8.02] | 4.00 [3.00 to 4.02] | 3.50 [1.50 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 3.02]

14. Secondary Outcome: Part A: Apparent Terminal Elimination Half-life (t1/2)
Description: Apparent terminal elimination half-life following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
hours | 18.5 (12.0) | 15.0 (27.4) | 15.7 (22.9) | 18.1 (29.3) | 17.6 (11.1) | 16.4 (12.1) | 14.8 (14.0)

15. Secondary Outcome: Part A: Apparent Total Clearance (CL/F)
Description: Apparent total clearance following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
liters per hour | 4.76 (18.8) | 5.00 (43.2) | 4.94 (36.9) | 4.74 (18.0) | 4.89 (28.3) | 4.61 (23.9) | 5.52 (17.9)

16. Secondary Outcome: Part A: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Description: Apparent volume of distribution during the terminal phase following single oral dose of KRP-A218
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male)
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 6 | 6
liters | 127 (16.4) | 108 (26.9) | 112 (14.2) | 124 (37.4) | 124 (31.5) | 109 (30.3) | 117 (20.2)

17. Secondary Outcome: Part B: Area Under the Concentration-time Curve Over a Dosing Interval (AUC0-τ)
Description: Assessment of the area under the concentration-time curve over a dosing interval (AUC0-τ)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL
  Day 1 | 254 (13.7) | 560 (18.7) | 1170 (38.8) | 1760 (27.5)
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 395 (24.1) | 813 (24.5) | 1630 (21.9) | 2760 (35.0)
Statistical Analysis 1: Comparison: Part B: 2 mg KRP-A218 vs Part B: 4 mg KRP-A218 vs Part B: 8 mg KRP-A218 vs Part B: 11 mg KRP-A218; Dose Proportionality Assessment. KRP-A218 assessed across the following dose levels: 2 mg, 4 mg, 8 mg, and 11 mg. Dose proportionality results for Part B are only for the Day 14 profile (not Day 1); Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Slope = 1.11, 95% CI 2-sided [0.966 to 1.26] — Between-subject geometric coefficient of variation was 26.9. Data were analyzed using a power model

18. Secondary Outcome: Part B: Area Under Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-infinity)
Description: Assessment of the area under concentration-time curve from time 0 extrapolated to infinity (AUC0-infinity)
Time Frame: Day 1
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL | 367 (18.5) | 800 (24.2) | 1590 (42.5) | 2480 (34.2)

19. Secondary Outcome: Part B: Area Under Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast)
Description: Assessment of the area under curve from time 0 to the time of the last quantifiable concentration (AUC0-tlast)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL
  Day 1 | 253 (13.7) | 558 (18.7) | 1170 (38.8) | 1750 (27.5)
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 575 (28.2) | 1170 (29.1) | 2370 (24.7) | 4050 (43.2)
Statistical Analysis 1: Comparison: Part B: 2 mg KRP-A218 vs Part B: 4 mg KRP-A218 vs Part B: 8 mg KRP-A218 vs Part B: 11 mg KRP-A218; [analysis description as in outcome 17, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Slope = 1.12, 95% CI 2-sided [0.945 to 1.29] — Between-subject geometric coefficient of variation was 32.1. Data were analyzed using a power model

20. Secondary Outcome: Part B: Maximum Observed Concentration (Cmax)
Description: Assessment of the maximum observed concentration (Cmax)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL
  Day 1 | 20.0 (14.2) | 44.0 (14.5) | 99.0 (32.4) | 137 (24.5)
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 29.9 (20.8) | 60.9 (23.5) | 121 (17.7) | 204 (28.8)
Statistical Analysis 1: Comparison: Part B: 2 mg KRP-A218 vs Part B: 4 mg KRP-A218 vs Part B: 8 mg KRP-A218 vs Part B: 11 mg KRP-A218; [analysis description as in outcome 17, analysis 1]; Test type: Equivalence — Study was not powered and confidence intervals were assessed for containing unity (1) within them; Slope = 1.10, 95% CI 2-sided [0.971 to 1.23] — Between-subject geometric of coefficient variation was 23.2. Data were analyzed using a power model

21. Secondary Outcome: Part B: Minimum Observed Concentration (Cmin)
Description: Assessment of the minimum observed concentration (Cmin)
Time Frame: Day 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 7 | 8
ng/mL | 9.09 (33.1) | 18.5 (35.3) | 33.0 (27.9) | 59.6 (45.1)

22. Secondary Outcome: Part B: Time of the Maximum Observed Concentration (Tmax)
Description: Assessment of the time of the maximum observed concentration (Tmax)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Median (Full Range); unit: hours
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours
  Day 1 | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.00 [2.00 to 4.00] | 3.50 [2.00 to 6.00]
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 3.00 [1.50 to 4.07] | 3.50 [2.00 to 4.00] | 4.00 [3.00 to 4.02] | 3.00 [1.50 to 3.00]

23. Secondary Outcome: Part B: Apparent Terminal Elimination Half-life (t1/2)
Description: Assessment of the apparent terminal elimination half-life (t1/2)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours
  Day 1 | 13.0 (18.8) | 12.5 (15.8) | 11.7 (12.4) | 12.6 (16.9)
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 18.8 (39.5) | 16.2 (22.1) | 17.6 (21.0) | 17.2 (20.5)

24. Secondary Outcome: Part B: Apparent Total Clearance (CL/F)
Description: Assessment of the apparent total clearance (CL/F)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
liters per hour
  Day 1 | 5.45 (18.5) | 5.00 (24.2) | 5.03 (42.5) | 4.44 (34.2)
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 5.06 (24.1) | 4.92 (24.5) | 4.90 (21.9) | 3.99 (35.0)

25. Secondary Outcome: Part B: Apparent Volume of Distribution During the Terminal Phase (Vz/F)
Description: Assessment of the apparent volume of distribution during the terminal phase (Vz/F)
Time Frame: Days 1 and 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 8 | 8
liters
  Day 1 | 102 (13.2) | 89.9 (13.8) | 84.6 (35.4) | 80.7 (24.0)
  Day 14: number analyzed (Participants) | 8 | 8 | 7 | 8
  Day 14 | 137 (52.1) | 115 (23.1) | 124 (34.1) | 99.0 (23.0)

26. Secondary Outcome: Part B: Observed Accumulation Ratio Based on Area Under the Concentration-Time Curve Over a Dosing Interval (ARAUC0-T)
Description: Observed accumulation ratio based on area under the concentration-time curve over a dosing interval (ARAUC0-T) in Part B
Time Frame: Day 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 7 | 8
ratio | 1.56 (13.6) | 1.45 (14.2) | 1.41 (19.1) | 1.57 (14.7)

27. Secondary Outcome: Part B: Observed Accumulation Ratio Based on Maximum Observed Concentration During the Dosing Interval (ARCmax)
Description: Observed accumulation ratio based on maximum observed concentration during the dosing interval (ARCmax) in Part B
Time Frame: Day 14
Population: Pharmacokinetic population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218
Number analyzed (Participants) | 8 | 8 | 7 | 8
ratio | 1.49 (14.0) | 1.38 (11.8) | 1.21 (17.0) | 1.49 (9.6)

28. Secondary Outcome: Part C: Number of Participants With Adverse Events
Description: as for outcome 1
Time Frame: Screening to follow-up (Approximately 7 weeks)
Population: Safety population
Measure: Number; unit: participants
Groups:
- Part C: Drug-drug Interaction Study: 200 mg Itraconazole Alone: Day 4: 2 × single oral doses of 200 mg itraconazole solution (10 mg/mL) administered with no additional water, approximately 12 hours apart, in the fasted state.
Arm/Group | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 200 mg Itraconazole Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
Number analyzed (Participants) | 12 | 12 | 12
participants
  Overall TEAEs | 5 | 3 | 6
  Serious TEAEs | 0 | 0 | 0
  TEAEs leading to discontinuation | 0 | 0 | 0
  TEAEs leading to death | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Over 4 months from screening (Days -28 to -2), throughout the treatment period (Days -1 to 72), and at follow-up (7 to 10 days postdose) if applicable.
Description: Fed/fasted group in Part A:
  * treatment-emergent adverse events (TEAEs) on/after Period 1, Day (D) 1 dose and prior to Period 2, D1 dose assigned to 3 mg KRP-A218 (Fasted Male)
  * TEAEs on/after Period 2, D1 dose assigned to 3 mg KRP-A218 (Fed Male)
  Part C:
  * TEAEs on/after D1 dose and prior to D4 dosing assigned to 1 mg KRP-A218
  * TEAEs on/after D4 dose and prior to D11 dosing assigned to 200 mg Itraconazole
  * TEAEs on/after D11 dose assigned to 1 mg KRP-A218 and 200 mg Itraconazole
Groups:
- Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone: Days 1 and 11: single oral dose of 1 mg KRP-A218 (with approximately 240 mL of room temperature water), in the fasted state.
- Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole: Days 5 to 13: single oral doses of 200 mg itraconazole, solution (10 mg/mL) administered with no additional water, in the fasted state.
Arm/Group | Part A: Placebo | Part A: 1 mg KRP-A218 (Fasted Male) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) | Part A: 3 mg KRP-A218 (Fasted Female) | Part A: 6 mg KRP-A218 (Fasted Male) | Part A: 12 mg KRP-A218 (Fasted Male) | Part A: 21 mg KRP-A218 (Fasted Male) | Part B: Placebo | Part B: 2 mg KRP-A218 | Part B: 4 mg KRP-A218 | Part B: 8 mg KRP-A218 | Part B: 11 mg KRP-A218 | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone | Part C: Drug-drug Interaction Study: 200 mg Itraconazole Alone | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8 | 0/8 | 0/8 | 0/8 | 0/8 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 3/5 | 4/6 | 3/6 | 2/6 | 2/6 | 3/6 | 2/6 | 6/8 | 3/8 | 7/8 | 5/8 | 5/8 | 5/12 | 3/12 | 6/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo (N=12) | Part A: 1 mg KRP-A218 (Fasted Male) (N=5) | Part A: 3 mg KRP-A218 (Fasted Male: Treatment Period 1) (N=6) | Part A: 3 mg KRP-A218 (Fed Male: Treatment Period 2) (N=6) | Part A: 3 mg KRP-A218 (Fasted Female) (N=6) | Part A: 6 mg KRP-A218 (Fasted Male) (N=6) | Part A: 12 mg KRP-A218 (Fasted Male) (N=6) | Part A: 21 mg KRP-A218 (Fasted Male) (N=6) | Part B: Placebo (N=8) | Part B: 2 mg KRP-A218 (N=8) | Part B: 4 mg KRP-A218 (N=8) | Part B: 8 mg KRP-A218 (N=8) | Part B: 11 mg KRP-A218 (N=8) | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 Alone (N=12) | Part C: Drug-drug Interaction Study: 200 mg Itraconazole Alone (N=12) | Part C: Drug-drug Interaction Study: 1 mg KRP-A218 + 200 mg Itraconazole (N=12)
Faeces soft (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 1 | 1 | 2 | 2 | 4 | 2 | 6 | 3 | 4 | 3 | 3 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dyschezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Catheter site bruise (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hunger (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bleeding time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal volume decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each party agrees that all confidential information of the disclosing part is and shall we the sole property of the disclosing party. Without prejudice to any Labcorp Property, all test information, results, data and records developed by Labcorp specifically as a result of performing the study and related to the test materials or sponsor information shall be the confidential information of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/00/NCT04908800/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT04908800/SAP_001.pdf